CLINICAL TRIAL: NCT06707922
Title: A Multicenter, Prospective, Follow-up Study to Evaluate the Long-term Benefits of Peginterferon Alpha-2b Injection Combined With TDF in Patients With Chronic Hepatitis B
Brief Title: A Follow-up Study of Peginterferon Alfa-2b Combined With TDF in Patients With Chronic Hepatitis B
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TB2111IFN
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Chronic Hepatitis B
Keywords: Peginterferon Alfa; Tenofovir Disoproxil Fumarate; Relapse; Retreatment
MeSH Terms: conditions — Hepatitis B, Chronic; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (No Intervention): Participants who have achieved functional cure at the time of completion of TB1901IFN will be included and followed up for 5 years without any intervention.
- Cohort 2 (Experimental): Participants with S antigen decrease≥1log and the S antigen level <100IU/ml at enrollment, or who with S antigen decrease ≥1.5log and the S antigen level <1500IU/ml after TB1901IFN treatment, will initially treated with 72-week pulse treatment of peginterferon in combination with TAF, and then followed up to 5 years.
  Interventions: Drug: Peginterferon α-2b Injection; Tenofovir Alafenamide Fumarate
- Cohort 3 (No Intervention): Except for those who already enrollment in Cohort 2, Participants with functional cure achievement will enroll in Cohort 3, and follow-up for 5 years without any study intervention.

INTERVENTIONS:
Drug: Peginterferon α-2b Injection; Tenofovir Alafenamide Fumarate — Peginterferon α-2b Injection, subcutaneous injection, once a week. Tenofovir Alafenamide Fumarate, Oral administration, once a day.
  Arms: Cohort 2

SUMMARY:
Studies have shown that chronic hepatitis B patients with low levels of HBsAg after nucleos(t)ide analog therapy have a higher chance of functional cure with sequential or combined pegylated interferon therapy, with about 30-50% of patients achieving HBsAg clearance and discontinuing therapy.

There are some clinical practices on the long-term benefits of discontinuing antiviral therapy, but there is a lack of evidence-based clinical studies, especially on the relapse rate, duration of relapse, and factors influencing relapse after achieving functional cure. Furthermore, there is no guideline or expert consensus on the follow-up management strategy for patients who haven't achieved functional cure but whose HBsAg levels have been substantially reduced by treatment and are at low levels.

Therefore, this study is planned to enroll participants who have completed the TB1901IFN to evaluate the long-term benefit of Peginterferon in combination with tenofovir disoproxil fumarate（TDF） and relapse in patients who have achieved functional cure, for participant with low-level HBsAg at the end of treatment, peginterferon combined with tenofovir alafenamide fumarate （TAF）therapy will be administered to explore the efficacy and safety of starting treatment after a period of drug discontinuation. Participants will be divided into 3 cohorts based on functional achievement and/or HBsAg levels after completion of TB1901IFN

ELIGIBILITY:
Inclusion Criteria:

* Participants who completion of the TB1901IFN study ("completion" is defined as completion of more than 80% of trial medications (including peginterferon alfa and tenofovir disoproxil fumarate), or meeting criteria for early discontinuation and completion of consolidation therapy, as well as completion of discontinuation follow-up and 24-week post-discontinuation visit);
* Voluntary enrollment, understand and sign the informed consent form.

For cohort 1 only; - Subjects who have achieved functional cure (defined as the disappearance of HBsAg at the completion of TB1901IFN, with or without the appearance of HBsAb);

For cohort 2 only:

* At the completion of TB1901IFN, the S antigen level has decreased by ≥1 log compared to the baseline, with an S antigen level of less than 100 IU/ml, or the S antigen level has decreased by ≥1.5 log compared to the baseline, with an S antigen level of less than 1500 IU/ml;
* Willing to accept the treatment of peginterferon combined with TAF;

For cohort 3 only:

- Participants who have not achieved functional cure upon completion of TB1901IFN (defined as HBsAg ≥ 0.05 IU/ml)；

Exclusion Criteria:

- Suspected or confirmed HCC patients.

For Cohort 2 only:

* Suspected or confirmed liver cirrhosis.
* Pregnant, breastfeeding women, or those who plan to conceive during the combined medication treatment period.
* Evidence of acute severe liver injury: e.g. ALT > 10 times of the upper limit of normal (ULN), or a significant increase in ALT accompanied by a significant increase in bilirubin;
* Evidence of decompensated liver disease: serum total bilirubin > 2ULN, serum albumin < 35 g/L, prothrombin time extended by more than 3 seconds beyond ULN, prothrombin activity < 60%; or a history of decompensated liver cirrhosis;
* Kidney disease: acute or chronic nephritis, renal insufficiency, nephrotic syndrome, etc., or serum creatinine > 1ULN;
* Neutrophil count < 1.5×10^9/L, platelet count < 90×10^9/L;
* Severe retinopathy or other severe ophthalmic diseases;
* Other conditions deemed by the investigator to be unsuitable for participation in the cohort 2.

For cohort 3 only:

- Participants who plan to enter Cohort 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of Hepatocellular Carcinoma(HCC). | 5 years after the completion of the TB1901IFN study.
The incidence all-cause mortality. | 5 years after the completion of the TB1901IFN study.
Relapse within 5 years of discontinuation in participants who achieved functional cure. | 5 years after the completion of the TB1901IFN study.
  Relapse was defined as the occurrence of two consecutive time, interval greater than one month, HBsAg≥0.05 IU/ml at any time during the follow-up period
Rate of functional cure of re-initiation of combination therapy after discontinued for more than 24 weeks in participants who had a favorable outcome on prior therapy and obtained low levels of S antigen. | After completing the 72-week combined re-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Guiqiang Wang, Ph.D, Principal Investigator — Peking University First Hospital
Locations (30):
- China (30):
  - Peking University First Hospital, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - The fifth medical center of PLA General Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital Central South University, Changsha
  - Public Health Clinical Center of Chengdu, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - Mengchao Hepatobiliary Hosipital of Fujian Medical University, Fuzhou
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Guangzhou Eighth People's Hospital, Guangzhou
  - The Third Affiliated Hospital,SUN YAT-SEN University, Guanzhou
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Huashan Hospital ,Fudan University, Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - The Sixth People's Hospital of Shenyang, Shenyang
  - Peiking University Shenzhen Hospital, Shenzhen
  - The Third People's Hospital of shenzhen, Shenzhen
  - The First Hospital of Shanxi Medical University, Taiyuan
  - First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin
  - Tianjin Third Central Hospital, Tianjin
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - Traditional Chinese Medical hospital of Xinjiang Uygur Autonomous Region, Ürümqi
  - Tongji Hospital,Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Tangdu Hospital,Air Force Medical University, Xi'an
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen
  - Yanbian University Hospital/Yanbian Hospital, Yanji
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No